CLINICAL TRIAL: NCT05515562
Title: Effects of IV Omadacycline on Gut Microbiome
Brief Title: Effects of Intravenous (IV) Omadacycline on Gut Microbiome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: University of Houston (Other); High Point University (Other); Paratek Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00081259
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-02

CONDITIONS: Microbial Colonization
Keywords: Gut Microbiome; Clostridioides difficile
MeSH Terms: conditions — Communicable Diseases | interventions — omadacycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intravenous (IV) Omadacycline (Experimental): All participants will receive 5 days of IV omadacycline followed by 5 days of oral omadacycline
  Interventions: Drug: Omadacycline Injection

INTERVENTIONS:
Drug: Omadacycline Injection — All participants will receive Intravenous (IV) omadacycline
  Other Names: Omadacycline oral

SUMMARY:
Given the clinical need to improve upon current antibiotic regimens for the treatment of C. difficile infection with a particular focus on the impact of therapies on gut microbiome, this study proposes to characterize the impact of Intravenous (IV) omadacycline on gut microbiome of healthy volunteers.

DETAILED DESCRIPTION:
The plan to enroll eight healthy volunteers between the ages of 18 and 40 years and without history of cardiovascular, gastrointestinal, hepatic, or renal disease to receive 5 days of intravenous omadacycline followed by 5 days of oral omadacycline. Stool and saliva samples will be collected at pre-specified times and analyzed to characterize the impact of IV omadacycline on gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years of age
* Willing and able to comply with all study procedures
* Considered healthy without history of cardiovascular, gastrointestinal, hepatic, or renal disease
* males or females - females of child bearing potential must agree to use a highly effective contraception during the study and for at least 7 days after the last dose of omadacycline

Exclusion Criteria:

* Consumed probiotics within 30 days before enrollment
* Consumed antibiotics within 90 days prior to enrollment
* Known hypersensitivity to omadacycline or tetracycline-class antibiotics
* pregnant or breastfeeding
* in the opinion of the investigator is experiencing signs or symptoms of acute illness that increase the risk of adverse effects from participating in the study
* previously participated in the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C Williamson, PharmD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie the results reported in this article, after deidentification
Supporting Information: Study Protocol
Time Frame: Beginning 6 months following article publication and ending 36 months following article publication
Access Criteria: Researchers who provide a methodologically sound proposal

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intravenous (IV) Omadacycline
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intravenous (IV) Omadacycline
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.875 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Phylum Level Mean Proportional Relative Abundance
Description: In general, the healthy volunteer analyses will assess changes in total and species-specific microbiota over time as well as changes in microbial diversity.
Time Frame: Day 30
Measure: Mean (Standard Deviation); unit: % gram positive (+) for phylum
Arm/Group | Intravenous (IV) Omadacycline
Number analyzed (Participants) | 8
% gram positive (+) for phylum
  Actinobacteriota | 0.167 (0.0622)
  Bacteroidota | 0.0271 (0.0314)
  Bacillota | 0.686 (0.114)
  Euryarchaeota | 0.0391 (0.103)
  Verrucomicrobiota | 0.0371 (0.0750)
  Proteobacteria | 0.0399 (0.0610)
  Other Phyla <2% | 0.00324 (0.00809)

2. Primary Outcome: Phylum Level Mean Proportional Relative Abundance
Description: as for outcome 1
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: % gram positive (+) for phylum
Arm/Group | Intravenous (IV) Omadacycline
Number analyzed (Participants) | 8
% gram positive (+) for phylum
  Actinobacteriota | 0.130 (0.0390)
  Bacteroidota | 0.0135 (0.0152)
  Bacillota | 0.779 (0.0879)
  Euryarchaeota | 0.0388 (0.0933)
  Verrucomicrobiota | 0.0173 (0.0227)
  Proteobacteria | 0.0205 (0.0342)
  Other Phyla <2% | 0.00110 (0.00190)

3. Primary Outcome: Phylum Level Mean Proportional Relative Abundance
Description: as for outcome 1
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: % gram positive (+) for phylum
Arm/Group | Intravenous (IV) Omadacycline
Number analyzed (Participants) | 8
% gram positive (+) for phylum
  Actinobacteriota | 0.225 (0.0469)
  Bacteroidota | 0.0507 (0.0812)
  Bacillota | 0.432 (0.0814)
  Euryarchaeota | 0 (0.0001)
  Verrucomicrobiota | 0.131 (0.106)
  Proteobacteria | 0.158 (0.141)
  Other Phyla <2% | 0.00310 (0.00407)

4. Primary Outcome: Phylum Level Mean Proportional Relative Abundance
Description: as for outcome 1
Time Frame: Day 10
Measure: Mean (Standard Deviation); unit: % gram positive (+) for phylum
Arm/Group | Intravenous (IV) Omadacycline
Number analyzed (Participants) | 8
% gram positive (+) for phylum
  Actinobacteriota | 0.198 (0.101)
  Bacteroidota | 0.0459 (0.0848)
  Bacillota | 0.246 (0.191)
  Euryarchaeota | 0.152 (0.262)
  Verrucomicrobiota | 0.210 (0.203)
  Proteobacteria | 0.147 (0.112)
  Other Phyla <2% | 0.00105 (0.00144)

5. Primary Outcome: Bacterial DNA Per Gram of Stool
Description: nanograms (ng) per gram of stool for bacterial DNA
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: 10^7 ng/g
Arm/Group | Intravenous (IV) Omadacycline
Number analyzed (Participants) | 8
10^7 ng/g
  Bacteroides thetaiotaomicron | 2.74 (6.11)
  Blautia coccoides | 608 (2.39)
  Clostridium leptum | 3.84 (1.73)
  Prevotella | 14.9 (46.6)
  Eubacteria | 2220 (953)
  Enterobacteriaceae | 1.42 (5.57)

6. Primary Outcome: Bacterial DNA Per Gram of Stool
Description: nanograms (ng) per gram of stool for bacterial DNA
Time Frame: During Therapy up to Day 6
Measure: Mean (Standard Deviation); unit: 10^7 ng/g
Arm/Group | Intravenous (IV) Omadacycline
Number analyzed (Participants) | 8
10^7 ng/g
  Bacteroides thetaiotaomicron | .954 (3.05)
  Blautia coccoides | 30.0 (22.9)
  Clostridium leptum | .0488 (.0553)
  Prevotella | 2.41 (22.8)
  Eubacteria | 197 (157)
  Enterobacteriaceae | 9.77 (31.5)

7. Primary Outcome: Bacterial DNA Per Gram of Stool
Description: nanograms (ng) per gram of stool for bacterial DNA
Time Frame: End of Therapy up to Day 10
Measure: Mean (Standard Deviation); unit: 10^7 ng/g
Arm/Group | Intravenous (IV) Omadacycline
Number analyzed (Participants) | 8
10^7 ng/g
  Bacteroides thetaiotaomicron | 0.849 (1.43)
  Blautia coccoides | 9.97 (14.7)
  Clostridium leptum | .0148 (.0130)
  Prevotella | 4.25 (7.30)
  Eubacteria | 103 (113)
  Enterobacteriaceae | 21.9 (37.4)

8. Primary Outcome: Order Level Mean Proportional Relative Abundance
Description: Order Level Mean Proportional Relative Abundance - Relative abundance % for order
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Relative abundance % for order
Arm/Group | Intravenous (IV) Omadacycline
Number analyzed (Participants) | 8
Relative abundance % for order
  p_Actinobacteriota o_Bifidobacteriales | 0.0349 (0.0265)
  p_Actinobacteriota o_Coriobacteriales | 0.0925 (0.0389)
  p_Bacteroidota o_Bacteroidales | 0.0135 (0.0152)
  p_Euryarchaeota o_Methanobacteriales | 0.0388 (0.0933)
  p_Bacillota o_Erysipelotrichales | 0.0693 (00622)
  p_Bacillota o_Lachnospirales | 0.417 (0.157)
  p_Bacillota o_Lactobacillales | 0.0429 (0.0273)
  p_Bacillota o_Oscillospirales | 0.188 (0.0883)
  p_Bacillota o_Peptostreptococcales- Tissierellales | 0.0213 (0.0109)
  p_Bacillota o_Veillonellales- Selenomonadales | 0.0107 (0.00754)
  p_Verrucomicrobiota o_Verrucomicrobiales | 0.0173 (0.0227)
  p_Proteobacteria o_Enterobacterales | 0.0204 (0.0342)
  Other Orders <2% | 0.0336 (0.0320)

9. Primary Outcome: Order Level Mean Proportional Relative Abundance
Description: Order Level Mean Proportional Relative Abundance - Relative abundance % for order
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: Relative abundance % for order
Arm/Group | Intravenous (IV) Omadacycline
Number analyzed (Participants) | 8
Relative abundance % for order
  p_Actinobacteriota o_Bifidobacteriales | 0.105 (0.0358)
  p_Actinobacteriota o_Coriobacteriales | 0.120 (0.0314)
  p_Bacteroidota o_Bacteroidales | 0.0507 (0.0812)
  p_Euryarchaeota o_Methanobacteriales | 0.000447 (0.0001)
  p_Bacillota o_Erysipelotrichales | 0.0148 (0.0143)
  p_Bacillota o_Lachnospirales | 0.204 (0.0845)
  p_Bacillota o_Lactobacillales | 0.0505 (0.0632)
  p_Bacillota o_Oscillospirales | 0.0653 (0.0507)
  p_Bacillota o_Peptostreptococcales- Tissierellales | 0.0163 (0.0161)
  p_Bacillota o_Veillonellales- Selenomonadales | 0.0685 (0.0881)
  p_Verrucomicrobiota o_Verrucomicrobiales | 0.131 (0.106)
  p_Proteobacteria o_Enterobacterales | 0.158 (0.141)
  Other Orders <2% | 0.0175 (0.0168)

10. Primary Outcome: Order Level Mean Proportional Relative Abundance
Description: Order Level Mean Proportional Relative Abundance - Relative abundance % for order
Time Frame: Day 10
Measure: Mean (Standard Deviation); unit: Relative abundance % for order
Arm/Group | Intravenous (IV) Omadacycline
Number analyzed (Participants) | 8
Relative abundance % for order
  p_Actinobacteriota o_Bifidobacteriales | 0.164 (0.0979)
  p_Actinobacteriota o_Coriobacteriales | 0.0324 (0.0368)
  p_Bacteroidota o_Bacteroidales | 0.0459 (0.0848)
  p_Euryarchaeota o_Methanobacteriales | 0.152 (0.262)
  p_Bacillota o_Erysipelotrichales | 0.229 (0.0546)
  p_Bacillota o_Lachnospirales | 0.0616 (0.0473)
  p_Bacillota o_Lactobacillales | 0.0128 (0.0104)
  p_Bacillota o_Oscillospirales | 0.0363 (0.0725)
  p_Bacillota o_Peptostreptococcales- Tissierellales | 0.0156 (0.0238)
  p_Bacillota o_Veillonellales- Selenomonadales | 0.0915 (0.142)
  p_Verrucomicrobiota o_Verrucomicrobiales | 0.210 (0.203)
  p_Proteobacteria o_Enterobacterales | 0.147 (0.112)
  Other Orders <2% | 0.00783 (0.00772)

11. Primary Outcome: Order Level Mean Proportional Relative Abundance
Description: Order Level Mean Proportional Relative Abundance - Relative abundance % for order
Time Frame: Day 30
Measure: Mean (Standard Deviation); unit: Relative abundance % for order
Arm/Group | Intravenous (IV) Omadacycline
Number analyzed (Participants) | 8
Relative abundance % for order
  p_Actinobacteriota o_Bifidobacteriales | 0.0880 (0.0515)
  p_Actinobacteriota o_Coriobacteriales | 0.0779 (0.0530)
  p_Bacteroidota o_Bacteroidales | 0.0270 (0.0313)
  p_Euryarchaeota o_Methanobacteriales | 0.0391 (0.103)
  p_Bacillota o_Erysipelotrichales | 0.0356 (0.0365)
  p_Bacillota o_Lachnospirales | 0.416 (0.169)
  p_Bacillota o_Lactobacillales | 0.0306 (0.0265)
  p_Bacillota o_Oscillospirales | 0.0971 (0.0941)
  p_Bacillota o_Peptostreptococcales- Tissierellales | 0.0271 (0.0197)
  p_Bacillota o_Veillonellales- Selenomonadales | 0.0657 (0.119)
  p_Verrucomicrobiota o_Verrucomicrobiales | 0.0371 (0.0750)
  p_Proteobacteria o_Enterobacterales | 0.0400 (0.0611)
  Other Orders <2% | 0.0186 (0.0198)

ADVERSE EVENTS:
Time Frame: 31 days
Arm/Group | Intravenous (IV) Omadacycline
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous (IV) Omadacycline (N=8)
Nausea (Gastrointestinal disorders) | 7 (7)
Abdominal Discomfort (Gastrointestinal disorders) | 2 (2)
Infusion arm discomfort (Skin and subcutaneous tissue disorders) | 3 (3)
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/62/NCT05515562/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/62/NCT05515562/ICF_001.pdf